CLINICAL TRIAL: NCT06476613
Title: Pilot Study- Permissive Hypotension After Cardiac Surgery
Brief Title: Permissive Hypotension After Cardiac Surgery
Acronym: PHACS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Asishana A Osho, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003142
Record Dates: First submitted 2024-06-07; First posted 2024-06-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Permissive hypotension Intervention (Experimental): In addition to the regular care provided to cardiac surgery patients, those in the permissive hypotension intervention arm will have a MAP target > 60mmHg.
  Interventions: Other: Permissive Hypotension
- Standard of Care (No Intervention): Patients randomized to the standard of care arm will receive the regular care provided to cardiac surgery patients.

INTERVENTIONS:
Other: Permissive Hypotension — Patients will be randomized in 1:1 fashion to either a) Permissive Hypotension (MAP target > 60mmHg) or b) Usual Care. The duration of the intervention will extend until the patient no longer needs vasopressors to maintain prespecified MAP.
  Arms: Permissive hypotension Intervention

SUMMARY:
The objective of this pilot randomized controlled trial is to demonstrate the feasibility of implementing a pragmatic clinical trial randomizing patients to permissive hypotension versus usual care and to determine the impact of permissive hypotension on vasopressor exposure, ICU length of stay, markers of end organ perfusion, and clinically relevant patient outcomes. The data collected from this pilot study will be used as preliminary data for study design and grant applications for a larger multicenter randomized controlled trial.

DETAILED DESCRIPTION:
The investigators will perform a single center, open-label, randomized controlled trial in patients admitted to the HCICU after cardiac surgery at MGH. Patients who are hypotensive (MAP < 65mmHg) and/or require vasopressor support to maintain a MAP ≥ 65mmHg during the first 24 hours of ICU admission will be eligible for randomization. Patients will be randomized in 1:1 fashion to either a) Permissive Hypotension (MAP target >60mmHg) or b) Usual Care. The duration of the intervention will extend until the patient no longer needs vasopressors to maintain prespecified MAP. Outcomes of interest include continuous hemodynamics (both recorded values from EHR as well as the arterial line waveform data), vasopressor exposure (as measured by maximum Vasopressor-Inotrope Score, mean Vasopressor-Inotrope Score, and duration of vasopressor use), lactate clearance, rates of atrial fibrillation, need for renal replacement therapy, ICU length of stay, survival to hospital discharge, cognitive state at discharge using Montreal Cognitive Assessment score. Additionally, the investigators will perform exploratory analyses using the continuous arterial line waveform data to evaluate for potential differences in arterial waveform morphologies between groups to help discern the hemodynamic impacts of permissive hypotension and to potentially identify subphenotypes who may derive greater benefit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Schedules for elective or non-emergent cardiac surgery

Exclusion Criteria:

* Arrival to the CICU with severe shock determined any of the following: Norepinephrine dose >20mcg/min, Epinephrine >3mcg/min, Dobutamine >2.5mcg/kg/min, Milrinone >0.2mcg/kg/min
* Rapidly increasing pressors within 60 mins of arrival.
* Significant prior renal dysfunction (CKD >4), hemodialysis dependence
* Cirrhosis
* A neuropathology diagnosis warranting blood pressure goal
* Pre-specified MAP goal as determined by clinical team
* Carotid stenosis (> 50%) or prior stroke
* Bleeding requiring return to the OR
* Need for mechanical circulatory support
* Heart and Lung transplantation
* Aortic dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
MAP in mmHg | Through study completion, an average of 2 to 3 days
  (Mean arterial pressure) measured in millimetres of mercury
Vasoactive-Inotropic Score for duration of pressor need | Through study completion, an average of 2 to 3 days
  Weighted sum of all administered vasopressor and inotropic medications and quantifies the amount of pharmacological support in patients

SECONDARY OUTCOMES:
ICU and hospital length of stay | Through study completion, an average of a week
  Total ICU and hospital length of stay following cardiac surgery
Duration of inotrope and vasopressor exposure | Through study completion, an average of 2 to 3 days
  Total duration of inotrope and vasopressor support required
Duration of end organ support | Through study completion, an average of 2 to 3 days
  Total duration for end organ support
Mortality | Through study completion, an average of a week
  Occurrence of death during study intervention
Cognitive function assessed using Montreal Cognitive Assessment (MOCA) | Through study completion, an average of a week
  Brief screening instrument for cognitive function
Tissue perfusion pressure via continuous arterial waveform monitoring | Through study completion, an average of 2 to 3 days
  Hemodynamic monitoring to ensure optimal tissue perfusion and oxygen delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koponen T, Karttunen J, Musialowicz T, Pietilainen L, Uusaro A, Lahtinen P. Vasoactive-inotropic score and the prediction of morbidity and mortality after cardiac surgery. Br J Anaesth. 2019 Apr;122(4):428-436. doi: 10.1016/j.bja.2018.12.019. Epub 2019 Feb 18. PMID 30857599
- [Background] Lamontagne F, Richards-Belle A, Thomas K, Harrison DA, Sadique MZ, Grieve RD, Camsooksai J, Darnell R, Gordon AC, Henry D, Hudson N, Mason AJ, Saull M, Whitman C, Young JD, Rowan KM, Mouncey PR; 65 trial investigators. Effect of Reduced Exposure to Vasopressors on 90-Day Mortality in Older Critically Ill Patients With Vasodilatory Hypotension: A Randomized Clinical Trial. JAMA. 2020 Mar 10;323(10):938-949. doi: 10.1001/jama.2020.0930. PMID 32049269
- [Background] Lamontagne F, Marshall JC, Adhikari NKJ. Permissive hypotension during shock resuscitation: equipoise in all patients? Intensive Care Med. 2018 Jan;44(1):87-90. doi: 10.1007/s00134-017-4849-2. Epub 2017 May 27. No abstract available. PMID 28551721
- [Background] Lamontagne F, Meade MO, Hebert PC, Asfar P, Lauzier F, Seely AJE, Day AG, Mehta S, Muscedere J, Bagshaw SM, Ferguson ND, Cook DJ, Kanji S, Turgeon AF, Herridge MS, Subramanian S, Lacroix J, Adhikari NKJ, Scales DC, Fox-Robichaud A, Skrobik Y, Whitlock RP, Green RS, Koo KKY, Tanguay T, Magder S, Heyland DK; Canadian Critical Care Trials Group.. Higher versus lower blood pressure targets for vasopressor therapy in shock: a multicentre pilot randomized controlled trial. Intensive Care Med. 2016 Apr;42(4):542-550. doi: 10.1007/s00134-016-4237-3. Epub 2016 Feb 18. PMID 26891677